CLINICAL TRIAL: NCT01603342
Title: A Pilot Study to Determine the Impact of Clopidogrel (Plavix®) on Bleeding Associated With Punch Biopsies in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7HAEM-1954
Record Dates: First submitted 2012-05-16; First posted 2012-05-22 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Haemostasis; Healthy
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- clopidogrel (Experimental)
  Interventions: Drug: clopidogrel
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: clopidogrel — Following a baseline punch biopsy, all subjects will then receive oral clopidogrel (Plavix®) over a period of approximately 3 to 4 days. Once the subject has successfully had 3 days of clopidogrel dosing, a second biopsy (B1) will be performed
  Arms: clopidogrel
Drug: placebo — Following a baseline punch biopsy, all subjects will then receive oral placebo over a period of approximately 3 to 4 days. Once the subject has successfully had 3 days of clopidogrel dosing, a second biopsy will be performed
  Arms: Placebo

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to determine the feasibility of demonstrating a quantifiable change from baseline in punch biopsy-induced bleeding durations and blood loss volumes in healthy subjects after receiving clopidogrel anti-platelet therapy.

ELIGIBILITY:
Inclusion Criteria:

* PT within normal laboratory range

Exclusion Criteria:

* The receipt of any investigational drug within 1 month prior to this trial
* Use of anti-coagulation or anti-platelet therapy-defined as vitamin K antagonists, platelet antagonists, heparin (or low molecular weight heparin), aspirin or NSAIDs within 30 days prior to trial
* African-American race
* Weight above or equal to 160 kg
* Recent diagnosis of any illness that would be present concomitant to trial period

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Bleeding duration measured in minutes | From onset of bleeding till the end of the bleeding

SECONDARY OUTCOMES:
Blood volume reported in millilitres | From onset of bleeding till the end of the bleeding
Adverse events, including special attention to bleeding complications | From day 0 to days 11-17
Change in coagulation-related parameters | From baseline to 15 minutes after biopsy B1

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neptune City, New Jersey, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com